CLINICAL TRIAL: NCT00406510
Title: Comparison of Frequency of Use of Optive and Systane
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 5283
Record Dates: First submitted 2006-11-30; First posted 2006-12-04 (Estimated); Last update posted 2007-06-01 (Estimated); Status verified 2007-05

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

INTERVENTIONS:
Drug: Optive, Systane

SUMMARY:
The purpose of this study is subjectively compare duration of action between Optive and Systane.

ELIGIBILITY:
Inclusion Criteria:

* Males or females > 18 years old
* Mild to moderate dry eye symptoms
* Score of at least 2 and no more than 4 on the SESOD at the initial screening visit
* Likely to complete all study visits and able to provide informed consent

Exclusion Criteria:

* Current use of topical cyclosporine
* Known contraindications to any study medication or ingredients
* Active ocular diseases or uncontrolled systemic disease (blepharitis patients that are actively being treated or disease that is uncontrollable)
* Ocular surgery within the past 3 months,
* Active ocular allergies

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Milton Hom, OD, Principal Investigator — Private Practice
Locations (1):
- Private Practice, Azusa, California, United States